CLINICAL TRIAL: NCT02715271
Title: Study of TB Lesions Obtained in Surgery: in Search of Best Biomarkers Correlating With TB Pathology, Clinical Features, MDR Cases and Prognostic
Brief Title: Study of TB Lesions Obtained in Therapeutical Surgery
Acronym: SH-TBL
Status: Completed | Type: Observational
Sponsor: Fundació Institut Germans Trias i Pujol (Other)
Collaborators: National Center for Tuberculosis and Lung Disease, Tbilisi, Georgia (Other)
Responsible Party: Principal Investigator, Cris Vilaplana, Senior Researcher at the Experimental Tuberculosis Unit, Fundació Institut Germans Trias i Pujol
Other Study IDs: SH-TBL-1
Record Dates: First submitted 2016-03-02; First posted 2016-03-22 (Estimated); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Tuberculosis; Thoracic Surgery; Tuberculosis, Pulmonary; Tuberculosis, Multidrug-Resistant
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary; Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — For the prospective substudy only:
  The following samples will be prospectively collected from patients undergoing therapeutical surgery:
  * Tissue samples from the TB lesions
  * plasma
  * whole blood for RNA studies
  * urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Retrospective cohort: Tuberculosis patients submitted to therapeutical surgery during the last 2-5 years.
  Interventions: Procedure: therapeutical surgery for TB
- Prospective cohort: Tuberculosis patients prospectively submitted to therapeutical surgery.
  Interventions: Procedure: therapeutical surgery for TB

INTERVENTIONS:
Procedure: therapeutical surgery for TB — Patients undergoing therapeutical surgery for tuberculosis (DS- and MDR/XDR-TB) indicated as per clinical routine

SUMMARY:
The correlation of the morphologic, microbiological, genetic and histopathological characteristics of TB lesions obtained in therapeutical surgery with the clinical forms and features of the patients will provide essential information

1. on the role of the host in the mechanisms associated to the generation and evolution of active TB and
2. about future diagnostic and/or prognostic biomarkers of TB disease. All this information could be used for patients stratification and/or to design new therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing therapeutical surgery for their Pulmonary Tuberculosis at NCTLD in Tbilisi, Georgia indicated as per clinical routine

Exclusion Criteria:

* Non consenting to donate samples and/or data for the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing therapeutical surgery for their Pulmonary Tuberculosis at NCTLD in Tbilisi, Georgia
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2016-09; Primary Completion 2024-05 (Actual); Study Completion 2024-05 (Actual)

PRIMARY OUTCOMES:
Description of Clinical and Epidemiological Data of the TB patients enrolled | at baseline
  for both the Retrospective and Prospective Substudies; descriptive analysis; data recorded in a spreadsheet created ad-hoc
Description of the Histopathological characteristics of the TB lesions of TB patients enrolled | at baseline
  for both the Retrospective and Prospective Substudies; descriptive analysis; data recorded in a spreadsheet created ad-hoc
Obtention of a genic-proteomic profile of TB lesions tissues which correlate to the histopathology of the granulomas and/or the clinic-pathological features of TB patients | at baseline
  only for Prospective Substudy; descriptive analysis, correlation with histopathological characteristics of TB lesions and with clinical and epidemiological data of TB patients

SECONDARY OUTCOMES:
Change in Immunological responses | at baseline; and at the moment of discharge, an average of at day 15 post-enrollment
  only for Prospective Substudy. Immunological responses will be measured 2.1.3. Identification of biomarkers in blood at protein level in blood and urine; validation in tissue and blood of genic biomarkers secreted (ELISA, qPCR, immunohistochemistry).
Change in Health Quality of Life Measurements | at baseline (before surgery) and through study completion, an average of 1 year
  measured with Health Quality of Life Questionnaires; only for Prospective Substudy

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Vilaplana, Dr, Principal Investigator — Fundació Institut Germans Trias i Pujol (IGTP)
Locations (1):
- National Center for Tuberculosis and Lung Diseases, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Data obtained will be openly available through Mendeley Data, under CC BY 4.0 license.
  Data set details:
  Vilaplana, Cristina; Vashakidze, Sergo; Gogishvili, Shota; Nikolaishvili , Keti; Despuig, Albert; Benito, Pau; Avramopoulos, Asimakis; García, Zaira; Téllez, Erica; Sarrias, Maria Rosa (2020), "SH-TBL project dataset", Mendeley Data, V1, doi: 10.17632/knhvdbjv3r.1
Time Frame: Once the results will be published.

REFERENCES:
- [Result] Vashakidze S, Despuig A, Gogishvili S, Nikolaishvili K, Shubladze N, Avaliani Z, Tukvadze N, Casals M, Cayla JA, Cardona PJ, Vilaplana C. Retrospective study of clinical and lesion characteristics of patients undergoing surgical treatment for Pulmonary Tuberculosis in Georgia. Int J Infect Dis. 2017 Mar;56:200-207. doi: 10.1016/j.ijid.2016.12.009. Epub 2016 Dec 19. PMID 28007659
- [Result] Benito P, Vashakidze S, Gogishvili S, Nikolaishvili K, Despuig A, Tukvadze N, Shubladze N, Avaliani Z, Vilaplana C. Impact of adjuvant therapeutic surgery on the health-related quality of life of pulmonary tuberculosis patients. ERJ Open Res. 2020 Aug 31;6(3):00083-2020. doi: 10.1183/23120541.00083-2020. eCollection 2020 Jul. PMID 32904577
- [Result] Moreira-Teixeira L, Stimpson PJ, Stavropoulos E, Hadebe S, Chakravarty P, Ioannou M, Aramburu IV, Herbert E, Priestnall SL, Suarez-Bonnet A, Sousa J, Fonseca KL, Wang Q, Vashakidze S, Rodriguez-Martinez P, Vilaplana C, Saraiva M, Papayannopoulos V, O'Garra A. Type I IFN exacerbates disease in tuberculosis-susceptible mice by inducing neutrophil-mediated lung inflammation and NETosis. Nat Commun. 2020 Nov 4;11(1):5566. doi: 10.1038/s41467-020-19412-6. PMID 33149141
- [Result] Fonseca KL, Maceiras AR, Matos R, Simoes-Costa L, Sousa J, Ca B, Barros L, Fernandes AI, Mereiter S, Reis R, Gomes J, Tapia G, Rodriguez-Martinez P, Martin-Cespedes M, Vashakidze S, Gogishvili S, Nikolaishvili K, Appelberg R, Gartner F, Rodrigues PNS, Vilaplana C, Reis CA, Magalhaes A, Saraiva M. Deficiency in the glycosyltransferase Gcnt1 increases susceptibility to tuberculosis through a mechanism involving neutrophils. Mucosal Immunol. 2020 Sep;13(5):836-848. doi: 10.1038/s41385-020-0277-7. Epub 2020 Mar 13. PMID 32203062
- [Derived] Moreno-Molina M, Shubladze N, Khurtsilava I, Avaliani Z, Bablishvili N, Torres-Puente M, Villamayor L, Gabrielian A, Rosenthal A, Vilaplana C, Gagneux S, Kempker RR, Vashakidze S, Comas I. Genomic analyses of Mycobacterium tuberculosis from human lung resections reveal a high frequency of polyclonal infections. Nat Commun. 2021 May 11;12(1):2716. doi: 10.1038/s41467-021-22705-z. PMID 33976135
- See also: website of the Experimental Tuberculosis Unit, Fundacio Institut Germans Trias i Pujol — http://unitatdetuberculosiexperimental.wordpress.com

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2016-04-20): https://cdn.clinicaltrials.gov/large-docs/71/NCT02715271/Prot_ICF_000.pdf